CLINICAL TRIAL: NCT00475150
Title: A Phase II Study of AZD2171 in the Treatment of Patients With Acute Leukemia and Myelodysplastic Syndrome.
Brief Title: Cediranib Maleate in Treating Patients With Relapsed, Refractory, or Untreated Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00129; NCI-2009-00129 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000544833; MCCRC-MC048H; MC048H (Other: Mayo Clinic); 7135 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH); NCT01646983 (obsolete NCT alias); NCT01664455 (obsolete NCT alias)
Record Dates: First submitted 2007-05-16; First posted 2007-05-17 (Estimated); Results first posted 2013-07-10 (Estimated); Last update posted 2017-02-15 (Actual); Status verified 2016-12

CONDITIONS: Adult Acute Myeloid Leukemia With 11q23 (MLL) Abnormalities; Adult Acute Myeloid Leukemia With Inv(16)(p13;q22); Adult Acute Myeloid Leukemia With t(15;17)(q22;q12); Adult Acute Myeloid Leukemia With t(16;16)(p13;q22); Adult Acute Myeloid Leukemia With t(8;21)(q22;q22); de Novo Myelodysplastic Syndromes; Previously Treated Myelodysplastic Syndromes; Recurrent Adult Acute Myeloid Leukemia; Secondary Acute Myeloid Leukemia; Secondary Myelodysplastic Syndromes; Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Congenital Abnormalities; Leukemia, Myeloid, Acute | interventions — cediranib

ARMS (1):
- Treatment (enzyme inhibitor therapy) (Experimental): Patients receive oral cediranib maleate QD on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cediranib maleate; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: cediranib maleate — Given orally
  Other Names: AZD2171; Recentin
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This phase II trial is studying how well cediranib maleate works in treating patients with relapsed, refractory, or untreated acute myeloid leukemia or high-risk myelodysplastic syndrome. Cediranib maleate may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth and by blocking blood flow to the cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the objective response rate in patients with relapsed, refractory, or untreated acute myeloid leukemia or high-risk myelodysplastic syndromes treated with AZD2171 (cediranib maleate).

SECONDARY OBJECTIVES:

I. Determine the toxicity of this drug in these patients. II. Determine the response duration, event-free survival, and overall survival of patients treated with this drug.

III. Determine the hematological response rate in patients treated with this drug.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (acute myeloid leukemia vs myelodysplastic syndromes).

Patients receive oral cediranib maleate once daily (QD) on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity. Patients undergo bone marrow biopsy at baseline and on day 28 for correlative studies. Samples are analyzed for circulating endothelial cells, VEGF receptor expression, and leukemic blasts via flow cytometry and microvessel density via histopathological techniques.

After completion of study treatment, patients are followed up at 3 months and then every 6 months for up to 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed acute myeloid leukemia (AML) ormyelodysplastic syndromes meeting 1 of the following criteria:

  * Relapsed AML meeting any of the following criteria:

    * Good-risk cytogenetics (inv[16], t[8;21], or t[15;17]) in second orgreater relapse

      * Patients with AML t(15;17) must have failed prior tretinoin and arsenic-containing regimens AND progressed orrelapsed within 12 months of therapy
    * In first or greater relapse
  * Resistant AML

    * Unable to achieve first complete remission after at least 2 inductionregimens
  * Untreated AML meeting any of the following criteria:

    * At least 60 years of age
    * Preceding MDS
  * MDS

    * International Prognosis Scoring System (IPSS) risk groupof intermediate-2 or higher
* Patients with relapsed disease after allogeneic hematopoietic stem cell transplantation (HSCT) must be off allimmunosuppressive medications for at least 30 days and have no symptoms orsigns of graft-vs-host disease
* No active CNS metastasis

  * Patients with clinical signs of CNS disease or a history of CNS diseasewithin the past 6 months are required to undergo lumbar puncture to excludeCNS involvement
* No symptomatic leukostasis or requirement for leukapheresis
* Not eligible for allogeneic HSCTAND no suitable donor at the time of study entry

  * Patients who areeligible for HSCT, informed of the option, and choose not to proceed to HSCTare allowed
* ECOG performance status (PS) 0-2 OR Karnofsky PS 60-100%
* Bilirubin normal
* AST and/or ALT ≤ 2.5 times upper limit of normal
* Creatinine normal OR creatinine clearance ≥ 60 mL/min
* No proteinuria ≥ 1+ on 2 consecutive urinalysis taken ≥ 1 week apart
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No HIV positivity
* LVEF ≥ 45% by echocardiography
* Mean QTc ≤ 500 msec (with Bazett's correction)
* No other significant ECG abnormality
* No history of familial long QT syndrome
* No disseminated intravascular coagulation
* No history of allergic reactions attributed to compounds of similar chemical orbiological composition to AZD2171
* No concurrent uncontrolled illness, including, but not limited to, any of the following:

  * Hypertension
  * Thyroid disease
  * Ongoing or active infection
  * Symptomatic congestive heartfailure
  * Unstable angina pectoris
  * Cardiac arrhythmia
  * NYHA class III-IV heart disease

    * NYHA class II heart disease controlled with treatment allowed
  * Psychiatric illness or social situations that would limit study compliance
* See Disease Characteristics
* More than 4 weeks since prior chemotherapy (6 weeks fornitrosoureas or mitomycin C), radiotherapy, or major surgery and recovered

  * Hydroxyurea allowed to control peripheral blast count> 20,000/mcL prior to study entry and during the first 3 days of study therapy
* More than 4 weeks since prior and no concurrent growth factor or other cytokine support
* At least 30 days since prior investigational agents or participation in aninvestigational trial
* No more than 3 prior courses of induction chemotherapy

  * Induction chemotherapyis defined as that intended to induce complete remission and given at a time thatthe patient has active disease
* No concurrent CYP interactive medications
* No other concurrent investigational agents
* No concurrent drugs or biologics with proarrhythmic potential
* Prior and concurrent hydroxyurea allowed to control peripheral blast count> 20,000/mcL during the first 3 days of study therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2008-05; Primary Completion 2011-07 (Actual); Study Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Juckett, Principal Investigator — Mayo Clinic
Locations (5):
- United States (5):
  - Howard University Hospital, Washington D.C., District of Columbia
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Johns Hopkins University/Sidney Kimmel Comprehensive Cancer Center, Baltimore, Maryland
  - Wayne State University/Karmanos Cancer Institute, Detroit, Michigan
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between June 2008 and June 2011, 39 participants were accrued to this study.
Pre-assignment Details: A total of 23 AML (7 at 45 mg; 16 at 30 mg) and 16 MDS (all at 30 mg) were enrolled. The AML and MDS groups were analyzed for the primary endpoint separately.
Groups:
- Acute Myeloid Leukemia (AML); Myelodysplastic Syndrome (MDS): Patients receive 30 mg oral cediranib maleate QD on days 1-28. Treatment repeats every 28 days for up to 26 courses in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Started | 23 | 16
Completed | 23 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS) | Total
Number analyzed (Participants) | 23 | 16 | 39
Age, Continuous [Median (Full Range); unit: years] | 70 [61 to 86] | 73 [61 to 87] | 72 [61 to 87]
Gender [Count of Participants; unit: Participants]
  Female | 12 | 6 | 18
  Male | 11 | 10 | 21
Region of Enrollment [Number; unit: participants]
  United States | 23 | 16 | 39

OUTCOME MEASURES:

1. Primary Outcome: The Number of Confirmed Disease Response: Complete Response (CR), Partial Response (PR), and Hematologic Improvement (HI). A Confirmed Response is Defined to be an Objective Status of CR, PR, or HI Noted on 2 Consecutive Evaluations.
Description: Complete Response (CR) requires a repeat bone marrow with < 5% myeloblasts, hemoglobin ≥ 11 g/dl, neutrophils ≥ 1000/mm3, platelets ≥ 100,000/mm3, and no circulating blasts.
  Partial Response (PR) requires a bone marrow blast reduction of 50% or more, hemoglobin ≥ 11 g/dl, neutrophils ≥ 1000/mm3, platelets ≥ 100,000/mm3, and no circulating blasts.
  Hematologic Improvement (HI) requires one of the following:
  1. RBC transfusion independent participants are required to have >1.5 g/dL increase in hemoglobin,
  2. RBC transfusion-dependent participants are required to be transfusion independent,
  3. A 100% increase, and an absolute increase over 500mm^3 in Absolute Neutrophil Count,
  4. Participants with a pretreatment platelet count over 20,000/mm3 require an absolute increase of 30,000/mm^3 or more,
  5. Participants with platelet count below 20,000/mm3 require an increase over 20,000/mm^3 and by at least 100%.
Time Frame: At the end of cycles 1 and 3 and every 3 cycles thereafter up to 26 cycles
Population: All participants were evaluable for this endpoint.
Measure: Number; unit: participants
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 23 | 16
participants
  Complete Response (CR) | 0 | 0
  Partial Response (PR) | 0 | 0
  Hematologic Improvement | 0 | 1

2. Secondary Outcome: Overall Survival
Description: Defined as the time from date of registration to date of death due to any cause or date last known alive. The distribution of survival time will be estimated using the method of Kaplan-Meier.
Time Frame: Every cycle during treatment and every 6 months for up to 2 years after completion of study treatment
Population: All participants were evaluable for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 23 | 16
months | 3.71 [2.20 to 5.75] | 4.66 [1.97 to 10.81]

3. Secondary Outcome: Progression-free Survival
Description: Defined as the time from date of registration to date that disease progression was documented, death, or last date that progression-free status was documented, whichever comes first. Estimated using the method of Kaplan-Meier.
  Disease progression is defined as one of the following:
  * A ≥ 50% increase in bone marrow blasts from the best response, or
  * A 50% or greater decrement from maximum remission/response levels in neutrophils or platelets, or
  * A reduction in hemoglobin concentration by at least 1.5 g/dl, or
  * Transfusion dependence (without alternative explanation and sustained for at least 2 weeks).
Time Frame: Every 3 courses during treatment and then at 3 months and every 6 months for up to 2 years after completion of study treatment
Population: All participants are evaluable for this primary endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 23 | 16
months | 2.82 [1.15 to 5.35] | 4.30 [1.97 to 7.72]

4. Secondary Outcome: Duration of Response
Description: Measured from the time criteria are met for CR or PR (whichever is first recorded) until the first date that recurrent or progressive disease is objectively documented. Estimated using the method of Kaplan-Meier.
Time Frame: Every 3 courses up to 26 courses
Population: This endpoint was not analyzed due to lack of response.
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: The Number of Patients That Report Adverse Events Possibly, Probably, or Definitely Related to AZD2171.
Description: Graded using the Common Terminology Criteria for Adverse Events (CTCAE) version 3.0. All adverse events determined to be possibly, probably, or definately related to AZD2171 are included in this analysis.
Time Frame: Continuously during treatment up to 26 courses
Population: All participants were analyzed for this endpoint.
Measure: Number; unit: participants
Arm/Group | Acute Myeloid Leukemia (AML) | Myelodysplastic Syndrome (MDS)
Number analyzed (Participants) | 23 | 16
participants
  Grade 3 or Higher | 14 | 11
  Grade 4 or Higher | 7 | 5
  Grade 5 | 0 | 0

ADVERSE EVENTS:
Groups:
- All Patients Receiving Cediranib Maleate: All patients receiving oral cediranib maleate, regardless of diagnosis were analyzed for toxicity.
Arm/Group | All Patients Receiving Cediranib Maleate
Serious Adverse Events (participants affected / at risk) | 23/39
Other Adverse Events (participants affected / at risk) | 39/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving Cediranib Maleate (N=39)
Febrile neutropenia (Blood and lymphatic system disorders) | 2 (2)
Hemoglobin decreased (Blood and lymphatic system disorders) | 4 (6)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 1 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 2 (2)
Mucositis oral (Gastrointestinal disorders) | 1 (1)
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1 (1)
Fatigue (General disorders) | 7 (7)
Infection (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Sepsis (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (2)
INR increased (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (4)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 7 (10)
Platelet count decreased (Investigations) | 8 (10)
Weight loss (Investigations) | 1 (1)
Anorexia (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 2 (2)
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1 (1)
Intracranial hemorrhage (Nervous system disorders) | 1 (1)
Bladder hemorrhage (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Petechiae (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
Hypotension (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Patients Receiving Cediranib Maleate (N=39)
Hemoglobin decreased (Blood and lymphatic system disorders) | 3 (3)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Left ventricular failure (Cardiac disorders) | 1 (1)
Hypothyroidism (Endocrine disorders) | 2 (3)
Constipation (Gastrointestinal disorders) | 6 (6)
Diarrhea (Gastrointestinal disorders) | 21 (49)
Dry mouth (Gastrointestinal disorders) | 1 (1)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 2 (2)
Lower gastrointestinal hemorrhage (Gastrointestinal disorders) | 4 (4)
Mucositis oral (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 16 (22)
Oral pain (Gastrointestinal disorders) | 1 (1)
Rectal pain (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 5 (9)
Edema limbs (General disorders) | 5 (7)
Fatigue (General disorders) | 35 (66)
Bladder infection (Infections and infestations) | 1 (1)
Colitis, infectious (e.g., Clostridium difficile) (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (2)
Upper respiratory infection (Infections and infestations) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1)
Bruising (Injury, poisoning and procedural complications) | 4 (4)
Alanine aminotransferase increased (Investigations) | 1 (3)
Alkaline phosphatase increased (Investigations) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1)
Bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 2 (4)
INR increased (Investigations) | 1 (2)
Laboratory test abnormal (Investigations) | 1 (1)
Leukocyte count decreased (Investigations) | 3 (3)
Neutrophil count decreased (Investigations) | 12 (18)
Platelet count decreased (Investigations) | 19 (36)
Weight loss (Investigations) | 13 (23)
Anorexia (Metabolism and nutrition disorders) | 7 (9)
Blood glucose increased (Metabolism and nutrition disorders) | 3 (7)
Dehydration (Metabolism and nutrition disorders) | 1 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (3)
Bone pain (Musculoskeletal and connective tissue disorders) | 2 (5)
Chest wall pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Joint pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle weakness (Musculoskeletal and connective tissue disorders) | 11 (16)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 11 (15)
Headache (Nervous system disorders) | 10 (15)
Peripheral sensory neuropathy (Nervous system disorders) | 3 (6)
Hemorrhage urinary tract (Renal and urinary disorders) | 1 (1)
Protein urine positive (Renal and urinary disorders) | 19 (26)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 (2)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 27 (56)
Hemorrhage nasal (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 8 (13)
Dry skin (Skin and subcutaneous tissue disorders) | 1 (2)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 25 (40)
Hypotension (Vascular disorders) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less